CLINICAL TRIAL: NCT02571257
Title: An 8-Week, Double-Blind, Placebo-Controlled, Randomized, Multicenter Study in Hypercholesterolemic Patients to Determine the Efficacy and Safety of Combination Therapy With CI-1027 and a Statin
Brief Title: Efficacy and Safety of Gemcabene in Hypercholesterolemic Patients on Stable Statin Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1027-018
Record Dates: First submitted 2015-10-05; First posted 2015-10-08 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Hypercholesterolemia
Keywords: LDL-C; Lipid Regulator
MeSH Terms: conditions — Hypercholesterolemia | interventions — gemcabene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo treatment on stable background statin therapy
  Interventions: Drug: Placebo
- Gemcabene 300 mg QD (Experimental): Gemcabene (also known as CI-1027) treatment on stable background statin therapy
  Interventions: Drug: Gemcabene
- Gemcabene 900 mg QD (Experimental): Gemcabene (also known as CI-1027) treatment on stable background statin therapy
  Interventions: Drug: Gemcabene

INTERVENTIONS:
Drug: Gemcabene — 1-300 mg tablet, QD, 56 days
  Arms: Gemcabene 300 mg QD
Drug: Gemcabene — 3-300 mg tablets, QD, 56 days
  Arms: Gemcabene 900 mg QD
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of gemcabene on LDL-C and other lipid parameters in hypercholesterolemic patients on a stable dose of a statin.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females
* 18 to 65 years of age
* Baseline LDL-C ≥ 130 mg/dL (3.4 mmol/L)

Exclusion Criteria:

* If female, postmenopausal or surgically menopausal
* Triglycerides (TG) >400 mg/dL
* Creatine phosphokinase (CPK) >3 × the upper limit of normal (ULN)
* Body Mass Index (BMI) >35 kg/m2
* Uncontrolled diabetes mellitus (HbA1c >10%)
* Renal dysfunction (blood urea nitrogen [BUN] or creatinine >2 × ULN)
* Hepatic dysfunction (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] >2 × ULN)
* Myocardial infarction, severe or unstable angina pectoris, coronary angioplasty, coronary artery bypass graft, or any other major cardiovascular event resulting in hospitalization in previous month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2000-08; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
LDL-C - percent change from baseline at Week 8 | 56 days

SECONDARY OUTCOMES:
Plasma lipid levels - percent change from baseline at Week 8 | 56 days
  apolipoprotein B (apoB), total cholesterol (TC), C reactive protein (CRP), triglyceride (TG), very low density lipoprotein (VLDL-C), high density lipoprotein (HDL-C)
Adverse Events | 56 days
Clinical Laboratory | 56 days

REFERENCES:
- [Derived] Stein E, Bays H, Koren M, Bakker-Arkema R, Bisgaier C. Efficacy and safety of gemcabene as add-on to stable statin therapy in hypercholesterolemic patients. J Clin Lipidol. 2016 Sep-Oct;10(5):1212-22. doi: 10.1016/j.jacl.2016.08.002. Epub 2016 Aug 10. PMID 27678439